CLINICAL TRIAL: NCT01060410
Title: Exploration of Genetic Polymorphisms Related to Individual Variations of Side Effects of Cyclophosphamide in Systemic Lupus Erythematosus Treatment
Brief Title: Exploration of Genotype Based Personalized Prescription of Cyclophosphamide in Systemic Lupus Erythematosus Treatment
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Wenying Shu, Ph.D., Sun Yat-sen University
Other Study IDs: 30873124-CTX2008
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Lupus Erythematosus, Systemic; Adverse Effects
Keywords: Myelosuppression; Infection; Nausea
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Infections; Nausea | interventions — Amplified Fragment Length Polymorphism Analysis; Cyclophosphamide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction as well as for pharmacokinetic studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cyclophosphamide,low dose,continuous
  Interventions: Genetic: Polymorphism Analysis; Drug: Cyclophosphamide; Other: Pharmacokinetic analysis

INTERVENTIONS:
Genetic: Polymorphism Analysis — Analysis of genetic polymorphisms of the drug metabolic enzymes involving in the bio-activation and elimination of cyclophosphamide
Drug: Cyclophosphamide — intravenous injection, 0.2g, once every two days
Other: Pharmacokinetic analysis — laboratory analysis of concentration of cyclophosphamide and 4-OH-cyclophosphamide in plasma

SUMMARY:
The purpose of this study is to investigate the relationship between the side effects of cyclophosphamide in the treatment of systemic lupus erythematosus (SLE) in Han Chinese and the genetic polymorphisms of drug metabolizing enzymes and pharmacokinetics of cyclophosphamide.

DETAILED DESCRIPTION:
Cyclophosphamide is a widely applied agent in treatment of systemic lupus erythematosus. As an alkylating agent, cyclophosphamide is able to induce several side effects, including thinned hair, loss of appetite, nausea, vomiting, infection, myelosuppression, etc. However, the remarkable variability of the reactions to the drug -- the incidence of side effect or the outcome of the treatment -- has been observed among patients. Cyclophosphamide is a pro-drug, which require some enzymes in the liver to transform it into an active chemical to arouse alkylating function. And then it undergoes a series of detoxification steps catalyzed by the specific metabolic enzymes. This study is designed to explore the genetic variation among individuals in the key processes of the activation and elimination of cyclophosphamide in order to find out whether these genetic factors are associated to the side effects or efficacy. The further understanding into the factors concerning on the drug might imply possible solution to minimize the incidence of side effects in patients of systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

1. The patients must have been diagnosed as SLE according to the American College of Rheumatology (ACR) criteria published in 1997.
2. The patients must sign the informed consent. And for the patients who are under 18 years old, both the signatures of their legal guardians and that of the patients are required on the written informed consent.
3. The patients are receiving the standard regimen of 0.2g cyclophosphamide given as intravenous injection once every two days.

Exclusion Criteria:

1. Pregnant women, women in breast-feeding period and the women who refuse to take contraception measures during treatment.
2. Patients with poor compliance.
3. Patients who are also diagnosed of cancer or who are receiving cyclophosphamide in treatment of cancer, or other anti-cancer therapy.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SLE patients receiving treatment with cyclophosphamide
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2010-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Min Huang, PhD., Study Chair — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Xueding Wang, PhD., Study Director — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Wenying Shu, PhD., Principal Investigator — Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, China; Xiuyan Yang, MD., Study Director — Department of Rheumatology, the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China; Liuqin Liang, MD., Principal Investigator — Department of Rheumatology, the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, China
Locations (1):
- Institute of Clinical Pharmacology, School of Pharmaceutical Sciences, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Systemic lupus erythematosus — http://ghr.nlm.nih.gov/glossary=systemiclupuserythematosus
- See also: Help Me Understand Genetics — http://ghr.nlm.nih.gov/handbook
- See also: Cytochrome P450 — http://ghr.nlm.nih.gov/glossary=cytochromep450
- See also: Cyclophosphamide — http://www.nlm.nih.gov/medlineplus/druginfo/meds/a682080.html
- See also: Understanding Drug Therapy and Managing Side Effects — http://www.leukemia-lymphoma.org/attachments/National/br_1171992654.pdf